CLINICAL TRIAL: NCT04380103
Title: A Phase I/II Study of Irinotecan, Oxaliplatin, Capecitabine (XELOXIRI) and Bevacizumab as a First-line Therapy for Patients With Metastatic Colorectal Cancer
Brief Title: A Phase I/II Study of XELOXIRI and Bevacizumab as First-line Treatment in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Lin Yang, professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2271
Record Dates: First submitted 2020-05-03; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Cancer; Colorectal Cancer; Colorectal Adenocarcinoma
Keywords: metastatic colorectal cancer; metastatic colorectal adenocarcinoma; XELOXIRI; bevacizumab
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XELOXIRI/Bevacizumab (Experimental): drugs: Irinotecan, Oxaliplatin, Capecitabine, Bevacizumab bevacizumab 5mg/kg on day1, irinotecan 150mg/m2 or 165mg/m2 on day1, oxaliplatin 85mg/m2 on day1 and capecitabine 1000mg/m2 twice a day on day1-7, administered every 2 week for 12 cycles, after 12 cycles, administer bevacizumab 5mg/kg on day 1 and capecitabine 1000mg/m2 twice a day on day1-7 as maintenance therapy.
  Interventions: Drug: XELOXIRI/Bevacizumab

INTERVENTIONS:
Drug: XELOXIRI/Bevacizumab — bevacizumab 5mg/kg on day1, irinotecan 150mg/m2 or 165mg/m2 on day1, oxaliplatin 85mg/m2 on day1 and capecitabine 1000mg/m2 twice a day on day1-7 repeated every 2 week for 12 cycles, after 12 cycles, bevacizumab 5mg/kg on day 1 and capecitabine 1000mg/m2 twice a day on day1-7 as maintenance therapy repeated every 2 week
  Other Names: Irinotecan, Oxaliplatin, Capecitabine, Bevacizumab

SUMMARY:
The phase I/II study was designed to evaluate if the regimen of Irinotecan, Oxaliplatin, Capecitabine (XELOXIRI) and Bevacizumab is a superior first-line option for patients with metastatic colorectal cancer(mCRC) in terms of safety and efficacy.

DETAILED DESCRIPTION:
Recent studies have shown that the triplet-drug regimen FOLFOXIRI (irinotecan/oxaliplatin/fluorouracil) can further improves survival benefit for patients with metastatic colorectal cancer(mCRC) compared to standard two-drug regimens in first-line therapy, especially when combined with bevacizumab. However, the increased toxicities of FOLFOXIRI limited its usage. Capecitabine demonstrates a superior efficacy and safety than fluorouracil, so we designed this trial to evaluate if the XELOXIRI plus bevacizumab can be a better alternative to FOLFOXIRI plus bevacizumab. The phase I study is to determine the safety and the recommended phase II dose (RP2D) of XELOXIRI plus Bevacizumab. In the phase II study, we aim to determine the efficacy of the regimen as first-line therapy for mCRC and explore potential molecular biomarkers (genomes, circulating tumor cell) for toxicity forecasting or efficacy monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic colorectal adenocarcinoma;
* Age 18-80 years old;
* Eastern Cooperation Oncology Group (ECOG) performance score(<2);
* At least one measurable lesion for disease assessment according to RECIST version 1.1;
* Able to take oral medications;
* Previous fluoropyrimidine-based adjuvant or neoadjuvant chemotherapy was allowed only when it ended ≥ 6 months before study enrollment;
* No previous therapy for mCRC;
* Adequate organ functions as assessed by the following laboratory requirements: Leukocytes≥3.0x109/L, absolute neutrophil count≥1.5x109/L, platelet count≥100x109/L, hemoglobin≥9g/dL; serum bilirubin≤1.5x the upper limit of normal(ULN);Alanine aminotransferase(ALT) and aspartate aminotransferase(AST)≤3x ULN; serum creatinine≤1.5x ULN; calculated creatinine clearance or 24 hour creatinine clearance ≥60ml/min.
* An expected survival of at least 3 months;
* Willingly provide written informed consent to study procedures.

Exclusion Criteria:

* Patients with dysphagia, active peptic ulcer, intestinal obstruction, active gastrointestinal bleeding, peptic perforation, malabsorption syndrome or uncontrolled intestinal inflammatory diseases;
* With a history of extensive enterotomy or pelvic radiation therapy; Suffering from grade 2 or higher symptomatic peripheral neuropathy according to National Cancer Institute Common Toxicity (NCI-CTC) criteria;
* Uncontrolled central nervous system metastasis, disseminated intravascular coagulation or active infection;
* With concurrent cancer distinct from colorectal adenocarcinoma except cured skin basal cell carcinoma and cervical carcinoma in situ;
* Undergone a major operation, open biopsy or major traumatic injury within 28 days before study enrollment or have potential to receive major operation during the trial;
* Received central venous access device within 2 days before study enrollment;
* Any kind of concurrent cardiac disease with clinical meanings, such as cardiovascular accident, myocardial infarction, thromboembolism or hemorrhage within 6 months before enrollment, congestive heart failure ≤New York Heart Association (NYHA) class 2 or uncontrolled hypertension.
* With positive urine protein and 24-hour urinary protein content>1g;
* Have a tendency of bleeding or clotting;
* With nasty open wounds, ulcers or fractures;
* Current or recent treatment of anticoagulants, antiplatelet agent or nonsteroidal anti-inflammatory drugs, while aspirin of daily dose less than 325mg is allowed.
* With any illness or medical conditions that may jeopardize the patient's compliance or interfere the analyses or judgements of study results;
* Pregnancy or lactation at the time of study entry;
* With fertility but refuse to contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2020-04-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
dose-limited toxicity (DLT) | up to 1 year
  dose limited toxicities are evaluated in the phase I study according to CTCAE v5.0 and reviewed through the phase I study completion
maximum tolerated dose (MTD) | up to 1 year
  MTD is determined according to the DLT in the phase I study
recommended phase 2 dose (RP2D) | up to 1 year
  RP2D is determined according to DLT and MTD in the phase 1 study
objective response rate (ORR) | up to 2 years
  ORR is defined as the proportion of patients achieving complete response or partial response

SECONDARY OUTCOMES:
Adverse events (AEs) | though study completion, an average of 2 years
  Adverse events assessments are computed and categorized according to the Common Toxicity Criteria of the National Cancer Institute, version 5.0
progression-free survival (PFS) | though study completion, an average of 2 years
  PFS is defined as the time from randomization to the earliest evidence of disease progression (per RECIST v1.1), or death from any cause
overall survival (OS) | up to 5 years
  OS is defined as the time from randomized to death from any cause or to last contact
disease control rate (DCR) | up to 2 years
  DCR is defined as the proportion of patients achieving complete response, partial response or having stable disease
duration of response (DOR) | though study completion, an average of 2 years
  DOR is defined as the length from the first response occured to disease progression
time to response (TTR) | up to 2 years
  TTR is defined as the length from randomization to the first response occured.
the surgical resection rate of patients with liver-only metastases | up to 2 years
  the percentage of patients with liver-only metastases undergoing surgical resections during the trial therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - National Center/Cancer Hospital, China Academy of Medical Science and Peking Union Medical College, Beijing
  - National Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing